CLINICAL TRIAL: NCT06948851
Title: Development of New Postoperative Intraretinal Cystoid Changes With Respect to Postsurgical Treatment Strategies After Vitrectomy With Membrane Peeling Due to Epiretinal Membranes
Brief Title: New Postoperative Intraretinal Cystoid Changes After Vitrectomy With Membrane Peeling Due to Epiretinal Membranes
Status: Active, not recruiting | Type: Observational
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department, Professor, Sponsor-Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: ICC
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epiretinal membranes (ERM) are a macular disorder leading to metamorphopsia and a decrease in visual acuity. Peeling of ERM during vitrectomy is, up to date, the only possible treatment option, opening chances for improvements of visual acuity and metamorphopsia. Occurrence of new intraretinal cystoid changes was described to be associated with a lower level of visual acuity after surgery, compared to patients, that never had intraretinal cystoid changes Aim of our study was to analyze development of new intraretinal cystoid changes after vitrectomy with membrane peeling with respect to postsurgical treatment strategies.

DETAILED DESCRIPTION:
Epiretinal membranes (ERM) are a macular disorder leading to metamorphopsia and a decrease in visual acuity. While ERM are rare among young people, they have prevalence rates of up to 30% in the age groups of 70 years or older. Peeling of ERM during vitrectomy is, up to date, the only possible treatment option, opening chances for improvements of visual acuity and metamorphopsia. Nevertheless, there is a risk for development of new intraretinal cystoid changes after peeling of ERM in about 10% of patients. Preoperative presence of intraretinal cystoid changes was already described as a risk factor for postsurgical presence of intraretinal cystoid changes and and occurrence of new intraretinal cystoid changes was described to be associated with a lower level of visual acuity after surgery, compared to patients, that never had intraretinal cystoid changes. Biomarker in presurgical optical coherence tomography (OCT) have been described to be associated with postsurgical results. Using a multivariable approach of analysis, presurgical DRIL and higher central macular thickness (CMT) were significant negative predictors on postsurgical visual acuity three months after surgery. However, influence of preoperative OCT biomarkers on development of new postsurgical intraretinal cystoid changes was not examined in theses studies. Aim of our study was to analyze development of new intraretinal cystoid changes after vitrectomy with membrane peeling with respect to postsurgical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* presence of an idiopathic ERM with decrease in visual acuity affecting activities of the daily life
* undergone pars plana vitrectomy with membrane peeling with application of periocular triamcinolone acetonide and a prolonged application of steroidal eye drops for three months after surgery, performed by a single surgeon in the time period from 01/08/2020 to 31/05/2023.
* presence of a follow-up examination at our department three months after surgery (+-1 month), including OCT with accurate image quality for analyzing the presence or absence of intraretinal cystoid changes and visual acuity testing.
* age of 18 years of older.

Exclusion Criteria:

* age below 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients having undergone pars plana vitrectomy with membrane peeling with application of periocular triamcinolone acetonide and a prolonged application of steroidal eye drops after surgery for at least 3 months. To examine differences in development of new postoperative cystoid changes outcomes will be compared with a historical group of patients, that did not receive periocular triamcinolone acetonide and had a postoperative application of steroidal eye drops for one month.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
new postoperative intraretinal cystoid changes | 3 months after surgery
  presence of new postoperative intraretinal cystoid changes is assessed from OCT images 3 months after surgery

SECONDARY OUTCOMES:
Maximum diameter of postoperative intraretinal cystoid changes | 3 months after surgery
  Maximum diameter is measured in µm from OCT images 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Leisser, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell P, Smith W, Chey T, Wang JJ, Chang A. Prevalence and associations of epiretinal membranes. The Blue Mountains Eye Study, Australia. Ophthalmology. 1997 Jun;104(6):1033-40. doi: 10.1016/s0161-6420(97)30190-0. PMID 9186446
- [Background] Bu SC, Kuijer R, Li XR, Hooymans JM, Los LI. Idiopathic epiretinal membrane. Retina. 2014 Dec;34(12):2317-35. doi: 10.1097/IAE.0000000000000349. PMID 25360790
- [Background] Frisina R, Pinackatt SJ, Sartore M, Monfardini A, Baldi A, Cesana BM, Semeraro F, Bratu A, Parolini B. Cystoid macular edema after pars plana vitrectomy for idiopathic epiretinal membrane. Graefes Arch Clin Exp Ophthalmol. 2015 Jan;253(1):47-56. doi: 10.1007/s00417-014-2655-x. Epub 2014 May 25. PMID 24859385
- [Background] Leisser C, Hirnschall N, Hackl C, Doller B, Varsits R, Ullrich M, Kefer K, Karl R, Findl O. Risk factors for postoperative intraretinal cystoid changes after peeling of idiopathic epiretinal membranes among patients randomized for balanced salt solution and air-tamponade. Acta Ophthalmol. 2018 Jun;96(4):e439-e444. doi: 10.1111/aos.13635. Epub 2018 Feb 20. PMID 29461674
- [Background] Leisser C, Amon DL, Huemer JC, Findl O. Diagnostic Reliability of Optical Coherence Tomography Biomarkers for Postsurgical Success in Visual Acuity in Patients with Idiopathic Epiretinal Membranes. Klin Monbl Augenheilkd. 2023 Oct;240(10):1207-1213. doi: 10.1055/a-1756-5243. Epub 2022 Apr 14. English, German. PMID 35426108